CLINICAL TRIAL: NCT00977834
Title: Assessment of Older Adults With Cancer: Feasibility of Computer Survey Methodology
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08147; P50CA107399-04 (NIH); K23AG026749-01 (NIH)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Assessment, Geriatric
Keywords: Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Patients with lymphoma or lung cancer
- Group 2: Caregivers

SUMMARY:
The purpose of this study is to evaluate the possibility of using a computer-based survey to gather information from older patients and their caregivers about the patient's daily activities, need for assistance, other medical problems, mood, nutrition and symptoms. Researchers will evaluate how many subjects are able to complete the survey on their own and the length of time needed to do so. Also, researchers will analyze the types of responses to each item and whether subjects are satisfied with the questionnaire.

DETAILED DESCRIPTION:
Patients older than age 65, in comparison to those younger than 65, have an 11-fold increased cancer incidence and a 16-fold increase in cancer mortality. The population at risk is growing rapidly: the number of adults age 65 and older is expected to double in the next 30 years. In order to adequately care for this growing population of older adults, oncologists need an assessment tool that provides information regarding an older individual's "functional age" in comparison to their "chronological age." The technology of geriatric assessment could potentially help identify those older adults who are more vulnerable to complications from cancer treatment. This inter-disciplinary assessment provides information regarding the patient's functional status, comorbid medical conditions, other medications, nutritional status, psychological state, social support, and cognition.

Hurria and colleagues developed a geriatric assessment for older adults with cancer, which includes well validated measures of functional status, comorbid medical conditions, nutritional status, psychological state, cognitive function, social activity, and social support. Pilot data demonstrates the feasibility of this assessment which can be completed in less than 30 minutes; however, this assessment is completed by "pencil and paper" and requires an interviewer to deliver and score the assessment.

Loscalzo, Clark, and colleagues have developed a computer methodology in order to assess the needs of patients with cancer of all ages. The assessment is completed by the patients and a scoring algorithm is developed to provide a summary of the patient's needs for the healthcare team. This assessment is highly successful at identifying the needs of patients of all ages.

In this protocol, we will merge the research interests of Hurria, Loscalzo, and Clark by developing a computer survey program to capture the physical and psychological needs of older adults with cancer. The goal of this study is to evaluate the feasibility of computer survey methodology among older adults with cancer. For the purposes of this protocol we will accrue patients with lymphoma and lung cancer.

Schema:

1. Identify an older adult (age 65 and older) with lymphoma or lung cancer.
2. Describe the study to the patient: patient consents or refuses.
3. Consenting patients complete the geriatric assessment via a computer survey.
4. The following feasibility data will be captured: length of time to complete the assessment, patient's need for assistance to complete the assessment, satisfaction with the use of computer survey methodology to complete the assessment.
5. The primary caretaker (if available) will be invited to participate in the protocol and complete a caregiver's survey of the patient's needs and questions about caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > age of 65
* Diagnosis of lymphoma or lung cancer
* Be able to provide informed consent

Exclusion Criteria:

* Not fluent in English (because not all questionnaires have been validated in other languages)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Brawerman Center-Outpatient Clinics (City of Hope)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering the geriatric assessment via computer survey methodology. | Upon enrollment (one timepoint)

SECONDARY OUTCOMES:
% of patients who do not enter the study and reason why | Upon enrollment (one timepoint)

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States